CLINICAL TRIAL: NCT03843164
Title: Lung Nodule Characterization by Artificial Intelligence Techniques
Acronym: CARANOD-IA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7311
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-02

CONDITIONS: Incidental Lung Nodule
Keywords: Solitary Pulmonary Nodule; Multidetector Computed Tomography; Artificial Intelligence
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Management of incidental lung nodule is difficult and mainly based on simple morphometric characteristics such as maximum size and shape. Radiomics could play a role in simplifying this management by orientating towards a benign or a malignant origin, by comparing advanced characteristics to a large database of lung nodules.

The primary purpose is to evaluate the performances of a novel tool based on radiomics to characterize incidental lung nodules, discovered on computed tomography.

The secondary objectives are:

* to evaluate the variation in the performances of the software based on various technical aspects of the CT, such as radiation dose, reconstruction algorithm, type of scanner,…
* to compare the performances of this software to those of expert readers,
* to analyze the potential impact of this software on patient's management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (at least 18 years old);
* With a chest CT acquired between Jan 1 2012 and Oct 1 2018 at the Strasbourg University Hospital;
* CT being available over the PACS and exhibiting at least one lung nodule;
* Patient having given its authorization for the exploitation of his medical data for this research.

Exclusion Criteria:

* Patient having expressed direct opposition to participation in this study;
* Patient under juridical protection;
* Patient under tutelage or guardianship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a chest CT acquired between Jan 1 2012 and Oct 1 2018 at the Strasbourg University Hospital;
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performances of a novel tool based on radiomics to characterize incidental lung nodules, discovered on computed tomography. | he period from January 1st, 2012 to October 01, 2018 will be examined
  The study concerns patients who performed a chest CT scan at Strasbourg University Hospitals between 01/01/2012 and 01/10/2018

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie B - NHC, Strasbourg, France